CLINICAL TRIAL: NCT03450096
Title: Continuous Lumbar Plexus Block Using Shamrock-technique for Postoperative Pain Treatment After Open Hip and Femoral Surgery in Children
Brief Title: Continous Lumbar Plexus Block in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too difficult to recruit patients
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPB in Children
Record Dates: First submitted 2018-02-16; First posted 2018-03-01 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Regional Anesthesia; Pediatric Anesthesia; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): A bolus injection for LPB of 0.5 ml/kg ropivacaine 3.75 mg/ml (max 40 ml will be performed and the catheter will be placed before surgical interventions. A continuous perineural infusion of 0.2 ml/kg/h ropivacaine 0.2%, starting immediately after initial bolus injection will be then administered
  Interventions: Other: LPB
- Control group (No Intervention): Patients in the control group (and in the active treatment group) will receive an opioid-based analgesia with a hydromorphone-patient controlled analgesia (PCA) depending on their analgesic demand

INTERVENTIONS:
Other: LPB — A bolus injection for LPB of 0.5 ml/kg ropivacaine 3.75 mg/ml (max 40 ml will be performed and the catheter will be placed before surgical interventions. A continuous perineural infusion of 0.2 ml/kg/h ropivacaine 0.2%, starting immediately after initial bolus injection will be then administered
  Arms: Treatment group

SUMMARY:
Randomised controlled prospective trial with 2 groups (active group with Lumbar plexus block (LPB)-catheter vs control group). In a randomized controlled trial, the investigators will investigate under controlled circumstances the effect of a LPB-catheter placed with ultrasound guided "Shamrock"-technique to improve postoperative pain treatment after unilateral open hip and femoral surgery in paediatric patients. The investigators will investigate the effect on opioid consumption and the reduction of opioid related side effects during the first 24 postoperative hours

DETAILED DESCRIPTION:
Paediatric patients undergoing orthopaedic surgery can experience severe pain in the postoperative period. When pain interferes with mobilization and joint movement, the rehabilitation phase is prolonged and painful. Approximately 13% of the children undergoing orthopaedic surgery report symptoms of chronic pain. Therefore, optimal pain treatment should be provided during and after the surgical procedure.

Intravenous opioids or continuous epidural blocks are commonly used for postoperative pain treatment after open hip and femoral surgery. However, side effects like nausea and vomiting, urinary retention, or pruritus are often related to these treatments.

Lumbar plexus blocks (LPB) are a safe and effective alternative for postoperative treatment after hip and femoral surgery. Single injection LPB techniques have shown to provide good pain relief during the early postoperative period in children. Paediatric patients might also benefit from a catheter technique giving a prolonged postoperative analgesia. LPB provide simultaneous sensory blocks of the femoral nerve and the obturator nerve. Both nerves are primarily responsible for the innervation to the femoral shaft, hip joint and the pelvic bones. In contrast to epidural anesthesia techniques, LPB has only unilateral effect. Patients therefore achieve higher mobilization levels, resulting in early rehabilitation.

Several ultrasound-guided lumbar plexus block techniques have been described in the past. The Shamrock technique is a new LPB-technique that has shown to improve visualization of the lumbar plexus, surrounding anatomy, and injection needle. The improved visualization can facilitate block performance and improve safety. A catheter technique will be used for LPB to provide prolonged postoperative analgesia.

In a randomized controlled trial, the investigators will investigate under controlled circumstances the effect of a LPB-catheter placed with ultrasound guided "Shamrock"-technique to improve postoperative pain treatment after unilateral open hip and femoral surgery in paediatric patients. The investigators will investigate the effect on opioid consumption and the reduction of opioid related side effects during the first 24 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients undergoing elective unilateral open hip and femoral surgery requiring general anaesthesia with intubation at the University Hospital - Inselspital in Bern.
* American Society of Anesthesiologist (ASA) physical status 1-3
* 8-16 year old with legal guardians providing written informed consent.

Exclusion Criteria:

* Obesity (BMI 30 kg/m2)
* Infeasibility to use a PCA pump
* Known or suspected infection of the skin at the site of needle puncture area
* Known allergy to ropivacaine
* Severe spine deformity
* Neuromuscular disease
* Coagulopathy.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption (in mg/kg) | 24 hours
  Cumulative opioid consumption (in mg/kg) in the first postoperative 24 hours in an active treatment group using LPB with a bolus of ropivacaine 0.375% and a continuous LPB-catheter infusion with ropivacaine 0.2 % compared with a control group without LPB

SECONDARY OUTCOMES:
Time to first opioid requirement | 4 hours
  Time to first opioid requirement
Total opioids consumption | up to 48 hours
  Total opioids consumption during 48 hours (in time periods 0-12 hours, 12-24 hours, 24-36 hours, and 36-48 hours)
Satisfaction of patients | 48 hours
  Satisfaction of patients measured via questionnaire
Occurrence of vomiting, nausea and pruritus | 48 hours
  Occurrence of vomiting, nausea and pruritus recorded in patient data management system

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Lehmann, PD Dr. med., Study Chair — Department Anesthesia and Pain Therapy, University Hospital Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No